CLINICAL TRIAL: NCT01695603
Title: Comparison of a New Automated Ventilatory Mode Named Intellivent to Standard Controlled Ventilation in Brain Injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Philippe Jolliet (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Prof. Philippe Jolliet, Main investigator, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Intellibrain
Record Dates: First submitted 2012-09-20; First posted 2012-09-28 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Brain Injured Patients
Keywords: Brain injury; Controlled ventilation; Intellivent; Capnia control
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard mode of controlled ventilation (No Intervention): Each brain injured patient will be ventilated during two hours with a standard mode of controlled ventilation.
- Intellivent arm (Experimental): Each brain injured patient will be ventilated during two hours with an automated mode of ventilation, the Intellivent mode.
  Interventions: Device: Intellivent

INTERVENTIONS:
Device: Intellivent
  Arms: Intellivent arm

SUMMARY:
Comparison of the ability of a new automated ventilatory mode named Intellibrain to maintain capnia and oxgen partial pressure within predefined ranges in comparison to the control of capnia and oxgen partial pressure obtained by using standard controlled ventilation modes in brain injured patients. Comparison of the numbers of alarms and required settings modifications observed with each ventilatory mode.

ELIGIBILITY:
Inclusion Criteria:

* Brain injury ( traumatic brain injury, subarachnoi8dal haemorrhage, intracerebral hemorrhage, ischemic stroke)
* Glasgow coma scale of 9 or less
* Controlled mechanical ventilation required
* Intracranial pressure monitoring required for clinical reasons

Exclusion Criteria:

* age under 16 years old
* clinical signs of brainstem lesions
* patients with withdrawal order or for whom organ donation is under discussion
* major haemodynamic instability
* High carbon dioxide alveoloarterial gradient (>10 mmHg) and/or suffering of severe hypoxemia (PaO2/FIO2 < 150 mmHg)
* Patients included in another interventional clinical study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Partial pressure of carbon dioxide
  The partial pressure of carbon dioxide (PaCO2) will be recorded every thirty minutes during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation

SECONDARY OUTCOMES:
Partial pressure of oxygen
  The partial pressure of oxygen (PaCO2) will be recorded every thirty minutes during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation
Number of alarms generated by the ventilator
  The number of alarms generated by the ventilator will be recorded during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation
Number of settings modifications
  The number of ventilator settings modifications required will be recorded during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation
Intracranial pressure
  Intracranial pressure will be recorded continuously during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation
Respiratory parameters
  Various respiratory parameters tidal volume, respiratory rate, minute ventilation, airway pressure) will be recorded during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation
Cerebral vasoreactivity
  Cerebral vasoreactivity will be studied from the intracranial pressure and invasive arterial pressure curves recorded during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation
Partial pressure of oxygen in the brain tissue if available
  Partial pressure of oxygen in the brain tissue, if available for clinical reasons, will be recorded during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation
Number of therapeutic actions needed to reduce intracranial pressure
  The number of therapeutic actions needed to reduce intracranial pressure will be recorded during two hours under standard controlled ventilation and during two hours under Intellivent ventilation.
Cerebral perfusion pressure
  Cerebral perfusion pressure will be recorded continuously during 2 hours under standard controlled ventilation and during 2 hours under Intellivent ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Jolliet, Prof, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Adult Intensive Care and Burn Unit, University hospital of Lausanne, Lausanne, Switzerland